CLINICAL TRIAL: NCT04915300
Title: Apabetalone for Pulmonary Arterial Hypertension: a Phase 2 Clinical Study
Brief Title: Apabetalone for Pulmonary Arterial Hypertension
Acronym: APPROACH-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Resverlogix Corp (Industry)
Responsible Party: Principal Investigator, Steeve Provencher, Professor, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-3625
Record Dates: First submitted 2021-05-19; First posted 2021-06-07 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Bromodomain-Containing Protein 4 (BRD4); Apabetalone; Pulmonary Arterial Hypertension; BRD4 inhibitor; Phase 2 clinical trial; Double-blind trial; Placebo-controlled trial
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — apabetalone

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apabetalone (Active Comparator): 100mg BID, 24-week (168±3 days) Treatment Period.
  Interventions: Drug: Apabetalone
- Placebo (Placebo Comparator): 24-week (168±3 days) period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apabetalone — Apabetalone 100mg p.o. (tablets) BID for 24 weeks treatment period.
  Arms: Apabetalone
Drug: Placebo — Placebo p.o. (tablets) BID for 24 weeks treatment period.
  Arms: Placebo

SUMMARY:
Throughout the past twenty years, numerous specific pharmacologic agents targeting the endothelial dysfunction associated with PAH have emerged. Short term placebo-controlled randomized trials assessing PAH-specific monotherapy with these molecules have reported improvements in pulmonary hemodynamics and exercise capacity. A recent meta-analysis also documented a reduction in short-term mortality of about ≈40% with such therapies. Several randomized clinical trials evaluating PAH-specific combination therapy have been conducted. Our recent meta-analysis showed that combination therapy was associated with a 35% risk reduction for the occurrence of clinical worsening compared to monotherapy. Nonetheless, the investigators also showed 17% of PAH patients receiving combination therapy still experienced clinical worsening over a median exposure of 16 weeks. Moreover, long-term survival on PAH-specific also therapy remains poor in the modern era, with a yearly mortality rate of 15 % in incident idiopathic PAH. The identification of innovative therapeutic targets and validation of these complementary therapeutic interventions are thus urgently needed in PAH.

The investigators and others (K. Stenmark, University of Colorado and H. Bogaard, VU University Medical Center, Amsterdam, personal communications), have published strong evidence that BRD4 plays a key role in the pathological phenotype in PAH accounting for disease progression and showed that BRD4 inhibition can reverse PAH in several animal models. Intriguingly, coronary artery disease (CAD) and metabolic syndrome are more prevalent in PAH compared with the global population, suggesting a link between these diseases. Interestingly, BRD4 is also a trigger for calcification and remodeling processes and regulates transcription of lipoprotein and inflammatory factors, all of which are important in PAH and CAD. Apabetalone, an orally available BRD4 inhibitor, is now in a clinical development stage with a good safety profile.

The overall objective of the study is to explore the efficacy and safety of apabetalone as an add-on therapy for adult PAH patients and to inform the conduct and the design of a Phase 3 trial.

The primary objective of the study is to assess the efficacy of apabetalone as evaluated by the change in PVR over a period of 24 weeks compared to placebo in adult subjects with PAH on stable background therapy.

Secondary objectives include changes at week 24 in 6MWD, plasma NT-proBNP concentration, WHO functional class, ESC/ERS risk stratification score, health-related quality of life and additional hemodynamic data from right heart.

Exploratory objectives are to evaluate the effects of apabetalone compared to placebo in adult subjects with PAH on mortality and clinically relevant morbidity events, and on circulating levels and transcription changes in whole blood markers of metabolism, vascular calcification, inflammation, DNA damage and leucocyte expression of BMPR2.

DETAILED DESCRIPTION:
This is a standard-design, double-blind, parallel-group, placebo-controlled trial.

Overall, 72 well-characterized PAH patients, 36 subjects in each treatment group (apabetalone 100 mg BID or matching placebo), that have been stable for >4 months on standard PAH-therapies, as per guidelines (Galie, Humbert et al. 2015) will be recruited in 8-15 participating centres (site selection currently ongoing). The participating centres will be recruited if they have the same approach to PAH patients in terms of choice and timing of treatments, and have expertise in performing trials in PAH. The initial Health Canada approval will be obtained. Apabetalone will be provided by Resverlogix Corp. Canada, but Resverlogix had no input into the trial design and will not be involved in the conduct of the trial, analysis, interpretation of the results or the final manuscript.

A 4-week pre-treatment phase will allow ensuring that patients are on stable doses of PAH medication. Patients will be given apabetalone 100mg BID or placebo.

Patients will be regularly followed to assess whether side effects. At baseline and week 24, a cardiac catheterization will assess changes in pulmonary hemodynamics and RV function.

An end-of-study visit is planned at week 28.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses.
3. Subject must be 18 to 75 years of age inclusive (18-80 years in case of PAH associated with scleroderma), at the time of signing the informed consent form.
4. PAH of idiopathic/hereditary/drug or toxin-induced origin; or associated with connective tissue diseases or simple congenital heart disease (atrial septal defect, ventricular septal defect, patent ductus arteriosus) corrected for >1 year;
5. Mean PA pressure >20mmHg, PVR >400 dyn.s.cm-5 with PA wedge pressure ≤15mmHg) and absence of acute vasoreactivity;
6. WHO functional class II or III;
7. Clinically stable with unchanged vasoactive therapy for ≥3 months;
8. Two 6MWD of ≥ 150m (the latter being used as baseline value);
9. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined as Absence of known liver cirrhosis, Haemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days, Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, Platelet count ≥ 100 x 109/L, Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN), Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 3.0 x institutional upper limit of normal and creatinine clearance estimated of ≥30 mL/min.
10. Patients must have a life expectancy ≥ 28 weeks.
11. Body mass index (BMI) within the range 18-40 kg/m2 (inclusive).
12. Patients of childbearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study treatment;
13. Patients must be postmenopausal, free from menses for >1 year, surgically sterilized, willing to use adequate contraception to prevent pregnancy, or agree to abstain from activities that could result in pregnancy; and agree to abstain lactating from enrollment through 3 months after the last dose of study treatment.
14. Male patients must use a condom during treatment and for 3 months after the last dose of apabetalone when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception (see appendix B for acceptable methods) if they are of childbearing potential.

Exclusion Criteria:

1. PAH related to HIV infection, portal hypertension;
2. Other types of pulmonary hypertension (Simonneau, Montani et al. 2019), including pulmonary related to left heart diseases, lung diseases, chronic thromboembolic disease or multifactorial mechanisms (PH groups 2-5, respectively);
3. Suspected pulmonary veno-occlusive disease;
4. A ventilation-perfusion lung scan or pulmonary angiography indicative of thromboembolic disease.
5. Significant restrictive (total lung capacity <70% predicted) or obstructive (FEV1/FVC<60% after a bronchodilator) lung disease;
6. DLCO <40%
7. Systolic blood pressure <90 mmHg;
8. Resting heart rate in the awake patient at rest <50 BPM or >110 BPM;
9. Acute RV failure or hospitalization within 30 days;
10. Received any investigational drug within 30 days;
11. Cardiopulmonary rehabilitation program planned or started ≤12 weeks prior to day 1;
12. Presence of ≥3 risk factors for heart failure with preserved ejection fraction, including:

    * BMI >30 kg/m2
    * Diabetes mellitus
    * Hypertension
    * Coronary artery disease
13. Recent cancer (<1yr, except for low grade and fully resolved non-melanoma skin cancer)
14. Recent bacterial infection (<30 days);
15. Anticipated survival less than 1 year due to concomitant disease.
16. Initiation of treatment with bosentan within 6 months (bosentan has been associated with a 5-10% risk or reversible raised in LFTs. This most commonly occurs within the first 6 months of treatment. Although there is no evidence of increased risk of apabetalone-related increases in LFTs amongst bosentan users, patients initiated on bosentan for <6 months will be excluded to minimize the risk of elevated LFTs falsely attributed to the study drug).
17. Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir). The required washout period prior to starting apabetalone is 2 weeks.*
18. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
19. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no.7).
20. Participation in another clinical study with an investigational product administered in the last 3 months
21. Patients with a known hypersensitivity to apabetalone or any of the excipients of their formulations.
22. Inability to consent
23. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
24. Breast feeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Placebo-corrected change from baseline in PVR at week 24 | Baseline, and 24 weeks later
  Right heart catheterization: Measuring PVR is performed in a standardized manner in catheterization laboratories of the participating centres, according to recommendations. Printed copies of waveforms will be kept for monitoring visits and documentation of the accuracy of the pressures and calculations.

SECONDARY OUTCOMES:
Changes at week 24 in 6MWD | Baseline, week 8 and week 24
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance (6 MWD) provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.
Changes at week 24 in plasma NT-proBNP concentration | Baseline, week 8 and week 24
Changes at week 24 in WHO functional class | Baseline, week 8 and week 24
  There are four functional classes that are used to rate how ill PH patients are. Class I: No symptoms of pulmonary arterial hypertension with exercise or at rest. Class II: No symptoms at rest but uncomfortable and short of breath with normal activity such as climbing a flight of stairs, grocery shopping, or making the bed. Class III: May not have symptoms at rest but activities greatly limited by shortness of breath, fatigue, or near fainting. Class IV: Symptoms at rest and severe symptoms with any activity.
Changes at week 24 in European Respiratory Society (ERS)/European Society of Cardiology (ESC) risk stratification score | Screening and Week 24
  The ERS/ESC risk stratification strategy will be used to categorize patients as low, intermediate or high risk. The cut-off values proposed in the guidelines will be graded 1-3 (1: low-, 2: intermediate- and 3: high-risk). For each patient, the sum of all grades will be divided by the number of variables and rounded to the next integer to define the risk group. The number of low-risk criteria per patients will also be assessed.
Change at week 24 in mean Pulmonary Artery Pressure (mPAP), mmHg obtained from right heart catheterization | Screening and Week 24
  The hemodynamic definition of pulmonary arterial hypertension (PAH) is a mean pulmonary artery pressure at rest greater than or equal to 25 mmHg in the presence of a pulmonary capillary wedge pressure less than or equal to 15 mmHg. These measurements can only be taken accurately during a right heart catheterization.
Change in cardiac output (L/min) | Screening and Week 24
  Catheterization
Change in right atrial pressure (RAP), mmHg | Screening and Week 24
  Catheterization
Change in mixed venous oxygen saturation (SvO2), % | Screening and Week 24
  Catheterization
Change at week 24 in HRQoL assessed using the EmPHasis-10 questionnaire | Screening and Week 24
  The Emphasis-10 questionnaire is a short questionnaire for assessing HRQoL in pulmonary arterial hypertension. It has excellent measurement properties and is sensitive to differences in relevant clinical parameters.

OTHER OUTCOMES:
Change in clinical worsening events | Baseline and Week 24
  Win ratio methodology will be used to evaluate the effects of apabetalone compared to placebo on mortality and clinically relevant morbidity events. The pairwise comparison proceeds in hierarchical fashion, using 1) all-cause mortality, followed by 2) frequency of PAH-related hospitalization; 3) a placebo-corrected change from baseline 6-minute walk distance >35 meters and; 4) a >20% relative placebo-corrected change in NTproBNP levels from baseline using the win ratio methodology. This method is based on the principle that each patient is compared with every other patient in a pairwise manner. This method gives a higher importance to all-cause mortality, followed by frequency of PAH-related hospitalization, exercise capacity and natriuretic peptide when patients cannot be differentiated on the basis of mortality, hospitalizations and functional status, respectively.
Circulating levels change in whole blood markers of metabolism | Baseline and Week 24
  Adiponectin, ApoA-I, LDL-C and HDL-C
Circulating levels change in whole blood markers of vascular calcification | Baseline and Week 24
  Alkaline phosphatase, osteoprotegerin, osteopontin, RUNX2
Circulating levels change in whole blood markers of inflammation | Baseline and Week 24
  C-reactive protein, fibrinogen, and inflammatory cytokines including IL-1 and IL-6
Circulating levels change in whole blood markers of DNA damage | Baseline and Week 24
  Comet assay, PARP1 expression
Change in PBMC expression of BMPR2 | Baseline and Week 24
  The proportion of patients with mutations in BMPR2 and key genes of the HR repair pathway

CONTACTS AND LOCATIONS:
Overall Officials: Steeve Provencher, MD, MSc, Principal Investigator — IUCPQ-UL; Pascale Blais-Lecours, PhD, Study Director — IUCPQ-UL
Locations (1):
- IUCPQ-UL, Québec, Canada

IPD SHARING:
Plan to Share IPD: No